CLINICAL TRIAL: NCT00011505
Title: Investigation of G-CSF-Induced Stem Cell Mobilization Potential in Patients With Diamond-Blackfan Anemia
Brief Title: Mobilization of Stem Cells With G-CSF for Collection From Patients With Diamond-Blackfan Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010097; 01-H-0097
Record Dates: First submitted 2001-02-22; First posted 2001-02-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-04

CONDITIONS: Diamond Blackfan Anemia
Keywords: G-CSF; Leukapheresis; Stem Cell Cryopreservation; Central Line Placement; G-CSF Administration; Stem Cell Preservation; Diamond Blackfan Anemia; Healthy Volunteer
MeSH Terms: conditions — Anemia, Diamond-Blackfan | interventions — Granulocyte Colony-Stimulating Factor; Leukapheresis

INTERVENTIONS:
Drug: G-CSF
Procedure: Leukapheresis

SUMMARY:
This study will provide information needed to develop more effective treatments for patients with Diamond-Blackfan anemia (DBA). Current treatments include steroids, such as prednisone, and blood transfusions. These treatments have potential long-term risk and side effects, including osteoporosis and impaired growth from steroids or iron overload from transfusions. In addition, as patients reach adulthood, they can develop acute leukemia or bone marrow failure. The only cure for DBA is bone marrow transplant, a procedure that itself carries serious risks and is an option for only about 25 percent of patients.

DBA is caused by a mutation (error) in a gene that codes for producing red blood cells from stem cells (blood-forming cells produced by the bone marrow). In 5 to 10 years, gene transfer therapy may prove to be an effective treatment for DBA. Before this treatment can be considered, however, more information is needed about DBA patients and how their stem cells function. This study will examine: 1) whether stem cells of patients with DBA respond to G-CSF the same way those of healthy people do. (G-CSF is a drug that causes stem cells to move from the bone marrow to the blood stream, where they can be collected more easily and in larger numbers by a procedure called leukapheresis, described below. If G-CSF does not work well in DBA patients, other collection strategies will have to be explored); and 2) whether the genetic error in DBA can be corrected by gene transfer into patients' stem cells.

Patients with Diamond-Blackfan anemia 4 years of age and older who weigh at least 27 pounds and who are dependent on red blood cell transfusions may be eligible for this study. Candidates will have a medical history taken and a physical examination and will be seen by the Clinical Center's Department of Medicine Transfusion for leukapheresis evaluation. They will have a bone marrow aspiration and biopsy to confirm the diagnosis of DBA. For these tests, the hip area is anesthetized and a needle is used to draw bone marrow from the hipbone. If needed, the procedure will be done under sedation.

Patients will be given G-CSF by injection under the skin for up to 6 days. Blood and stem cell counts will be measured from a teaspoon of blood drawn each morning. On the morning of the fifth dose, the patient will undergo leukapheresis for collection of stem cells. For this procedure, a large catheter (with a diameter no larger than that of a straw) is placed in an arm vein to allow blood to flow into a cell separator machine. Most children and some adults do not have veins large and strong enough for this tubing, so a large intravenous line called a "central line" is placed into a large vein in the neck or groin. This is done under sedation and with a local anesthetic. While the patient lies on a bed or recliner, whole blood is collected through a catheter in one arm or the central line, the stem cells are separated out by spinning, then the red cells, platelets and plasma are returned through a second catheter in the other arm or a second opening in the central line. The procedure takes about 3 to 5 hours, during which the patient can watch television or videos and have family members at the bedside for company. When the procedure is completed, the patient's participation in the protocol ends.

Some of the stem cells collected by leukapheresis will be used for research and some will be frozen and stored for possible future transplantation into the patient, if required.

DETAILED DESCRIPTION:
Diamond-Blackfan anemia (DBA) is a congenital hypoproliferative anemia that generally presents in infancy. The mainstays of treatment, prednisone and transfusion therapy, have long-term toxicity in many patients, and bone marrow transplantation with an HLA-matched donor is an option for only a minority of patients. Most importantly, patients with DBA have an increased risk of progression of myelodysplastic syndrome, leukemia, and aplastic anemia compared to the general population.

The characterization of potentially mutated genes in DBA is an area of active research, and at least one mutation present in about one-fourth of DBA patients may cause disease due to decreased production of a ribosomal protein. This finding raises the possibility that the disease, at least in some patients, may be correctable by genetic therapy, by which a normal copy of the mutated gene can be introduced into the "stem cells" which give rise to red cells.

It is therefore of interest to identify any particular characteristics of DBA patients which might delay or hinder the application of gene therapy to their disease. This pilot study of 15 patients is designed to evaluate: 1) the CD34+ cell mobilization response to administration of standard doses of granulocyte-colony stimulating factor (G-CSF), 2) the potential for stem cells from DBA patients to be collected by large volume leukapheresis of subjects who have been given G-CSF, and 3) the ability of these G-CSF mobilized cells to be transduced with vectors being developed for gene therapy applications. Outcome parameters to be monitored are the mobilization response to G-CSF, the safety profile and tolerance of G-CSF and leukapheresis, and the efficiency of transduction of DBA stem cells with standard gene therapy vectors. Effectiveness will be gauged by historical comparison of these parameters to normal healthy age-matched volunteer.

It is important to point out that there is no therapeutic intent to the majority of this protocol or direct benefit for enrolled patients. We do plan, however, to cryopreserve the remainder of the mobilized cells collected by apheresis for possible autologous transplantation in the event of the patient's progression to leukemia of bone marrow failure in the future.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female patients greater than or equal to 4 years of age and weighing at least 12 kg (27 lbs) will be included.

Diagnosis of DBA as defined by the onset of anemia before age 2; or, if after age 2, a positive family history of classical DBA or typical physical anomalies

Low reticulocyte counts (less than 30,000/ul)

Absent or blocked maturation of erythroid precursors in the bone marrow.

Red-cell transfusion dependence

Adequate birth control while on protocol

EXCLUSION CRITERIA:

Female patients that are pregnant or lactating

Neutrophil count less than 1000/uL or platelet count less than 100,000/uL

Positive DEB stimulation test

Evidence of transformation to MDS or AML on pre-study marrow aspiration and biopsy, or abnormal marrow cytogenetics.

History or evidence of clinically significant autoimmune inflammatory disease or significant cardiopulmonary disease by history or physical exam

Uncorrected coagulopathy

Renal disease (GFR less than 100mL/min/1/73 M(2)) as estimated for children by Schwartz formula. Adults (age greater than 21) excluded for serum Cr less than 2.5 mg/dL.

Hepatic disease (bilirubin greater than 2 mg/dL or transaminases greater than 7 times the upper limit of normal).

Seropositivity for hepatitis B (HbsAg), hepatitis C, or HIV will be excluded.

Other medical illness or condition which, in the opinion of the Investigators, may contraindicate participation in this study due to risk to patient or comprise of study integrity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2001-02; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kynaston JA, West NC, Reid MM. A regional experience of red cell aplasia. Eur J Pediatr. 1993 Apr;152(4):306-8. doi: 10.1007/BF01956739. PMID 8482277
- [Background] Ball SE, McGuckin CP, Jenkins G, Gordon-Smith EC. Diamond-Blackfan anaemia in the U.K.: analysis of 80 cases from a 20-year birth cohort. Br J Haematol. 1996 Sep;94(4):645-53. doi: 10.1046/j.1365-2141.1996.d01-1839.x. PMID 8826887
- [Background] Willig TN, Gazda H, Sieff CA. Diamond-Blackfan anemia. Curr Opin Hematol. 2000 Mar;7(2):85-94. doi: 10.1097/00062752-200003000-00003. PMID 10698294